CLINICAL TRIAL: NCT02035917
Title: Comparison of Tibial Plateau Fractures Outcomes Treated With Non-locking and Locking Plate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amin Nemati, Orthopedic surgery resident,Orthopedic department,Alzahra hospital,Isfahan University of Medical Sciences,Isfahan,Iran, Isfahan University of Medical Sciences
Purpose: Treatment
Other Study IDs: 392120
Record Dates: First submitted 2014-01-11; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Tibial Fracture
MeSH Terms: conditions — Tibial Fractures

ARMS (2):
- Locking plate (Experimental)
  Interventions: Device: Locking plate
- Non-Locking plate (Active Comparator)
  Interventions: Device: Non-Locking plate

INTERVENTIONS:
Device: Locking plate
  Arms: Locking plate
Device: Non-Locking plate
  Arms: Non-Locking plate

SUMMARY:
this study will perform to compare the results and functional outcomes of tibial plateau fractures treated with non-locking and locking plate fixation.

ELIGIBILITY:
Inclusion Criteria:

* unilateral closed tibia plateau fracture

Exclusion Criteria:

* patients who have been treated with casting or screw
* history of diabetes mellitus
* evidences of pathological fractures

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
knee society knee score | ten months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Tahririan, Orthopedic surgeon, Study Director — Department of Orthopedics, Kashani hospital, Isfahan University of Medical sciences, Isfahan, Iran; Mohsen Derakhshan, Orthopedic surgery resident, Principal Investigator — Department of Orthopedics, Kashani hospital, Isfahan University of Medical sciences, Isfahan, Iran
Locations (1):
- Vice Chancellery for Research of Isfahan University of Medical Sciences, Isfahan, Iran, Isfahan, Isfahan, Iran